CLINICAL TRIAL: NCT02577211
Title: Randomized Controlled Trial of Hypocaloric Hyperproteic Enteral Nutrition in the Critically Ill Patient
Brief Title: Hypocaloric Enteral Nutrition in the Critically Ill Patient
Acronym: hipoentnut
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lafrancol S.A. (Industry)
Collaborators: Hospital Universitario San Ignacio (Other); Pontificia Universidad Javeriana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: hnrct2
Record Dates: First submitted 2015-10-10; First posted 2015-10-16 (Estimated); Last update posted 2015-11-10 (Estimated); Status verified 2015-11

CONDITIONS: Critically Ill
Keywords: Critically ill; Enteral nutrition
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hipocaloric enteral nutrition (Experimental): 15 kcal per kg of body weight and 1.7 grams of protein per kg.
  Interventions: Dietary Supplement: Hipocaloric enteral nutrition
- Normocaloric enteral nutrition (Active Comparator): 25 kcal per kg of body weight and 1.7 grams of protein per kg.
  Interventions: Dietary Supplement: Normocaloric enteral nutrition

INTERVENTIONS:
Dietary Supplement: Hipocaloric enteral nutrition — 15 kcal/Kg of body weight
  Other Names: low caloric delivery
  Arms: Hipocaloric enteral nutrition
Dietary Supplement: Normocaloric enteral nutrition — 25 kcal/kg of body weight
  Arms: Normocaloric enteral nutrition

SUMMARY:
The aim of this study is to compare two nutritional regimes in critically ill patients. Patients will be randomized to standard care (25 kcal per kg) or to hypocaloric nutrition (15 kcal per kg). Both regimes will recive 1,7 g/Kg/dia The main outcome will be the SOFA (sequential organ failure assessment) score. The hypothesis is that hypocaloric hyperproteic diet decreases the incidence of organic failure in these patients.

DETAILED DESCRIPTION:
The research site will be the intensive care unit (ICU) of Hospital Universitario San Ignacio; eligible patients will >18 years of age with a presumed fasting period of at least 96 hours, with no contraindications for enteral nutrition. Patients with parenteral nutrition, pregnancy, diabetes, liver failure, renal failure, transplant protocol, or admitted from another hospital will be excluded. In all patients, the following information will be collected daily: enteral formula in ml, carbohydrate intake, insulin required (in IU), presence of hyper or hypoglicemia, presence of infections, among others.

The SOFA score will be assessed every two days until discharge from ICU.

ELIGIBILITY:
Inclusion Criteria:

* >18 years
* Estimated fasting period of at least 96 hours
* ICU patients

Exclusion Criteria:

* Parenteral nutrition
* Pregnancy
* Diabetes
* Liver failure
* Transplantation or in transplant protocol
* Previous nutrition support
* Chronic Renal failure

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2013-12; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Change in the intial SOFA (Sequential Organ Failure Assessment) score at 48 hours. | 48 hours after the onset of nutrition
  SOFA score evaluates six systems: respiratory, cardiovascular, coagulation, Central Nervous System, liver and renal. Each system gets a score from 0 (normal) to 4 (abnormal) and the sum of each score defines the final SOFA score, which 24 is the maximum score (high risk of morality) and 0 is the minimum score (low risk of mortality).

SECONDARY OUTCOMES:
Units of insulin require in a day | Within the first 4 days after the onset of nutrition
  This is an indirect measure of glycemic control, and is reported as a daily average of the units of insuline require in the first 4 days since nutritional regimen starts.
Number of days the patient requires mechanical ventilation. | Within the first 28 days after the onset of nutrition
  Measure daily
Number of days in the intensive care unit | Within the first 28 days after the onset of nutrition
  Measure daily
Mortality to 28 days | 28 days after the onset of nutrition
  We will interview each patient 28 days after the start of the study to assess the global mortality

CONTACTS AND LOCATIONS:
Overall Officials: Saul J Rugeles, MD, Principal Investigator — Hospital Universitario San Ignacio
Locations (1):
- Hospital Universitario San Ignacio, Bogotá, Bogota D.C., Colombia